CLINICAL TRIAL: NCT07302919
Title: Randomized, Double-Blind, Parallel, Controlled, Multicenter Study of Transarterial Chemoembolization (TACE) Plus ABCB1 Inhibition Versus TACE Alone in Patients With Hepatocellular Carcinoma: IMPACT-TACE
Brief Title: Transarterial Chemoembolization (TACE) Plus ABCB1 Inhibition Versus TACE Alone in Patients With Hepatocellular Carcinoma
Acronym: IMPACT-TACE
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-02072, bb24heim
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Hepato Cellular Carcinoma (HCC)
Keywords: Transarterial Chemoembolization (TACE)

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Parallel, Controlled, Multicenter Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental)
  Interventions: Combination Product: DEB-DoxNic-TACE
- Control Arm (Active Comparator)
  Interventions: Combination Product: current standard of care

INTERVENTIONS:
Combination Product: DEB-DoxNic-TACE — TACE (transarterial chemoembolization) with 1-3 mL drug-eluting beads (DEB) loaded with 33mg/ml doxorubicin (Dox) and 0.3mg/mL nicardipine (Nic)
  Arms: Experimental Arm
Combination Product: current standard of care — TACE (transarterial chemoembolization) with 1-3 mL drug-eluting beads loaded with 33mg/ml doxorubicin
  Arms: Control Arm

SUMMARY:
IMPACT-TACE is an investigator-initiated, prospective, multicenter, randomized, double-blinded, interventional trial to test the hypothesis that the simultaneous application of doxorubicin with the ABCB1 inhibitor nicardipine would significantly improve the success rate of TACE treatment.

DETAILED DESCRIPTION:
Liver cancer, also known as hepatocellular carcinoma (HCC), is the sixth most common tumor disease worldwide. It is an aggressive cancer that is very often fatal, as it is usually detected at a late stage when surgery is no longer possible. International guidelines recommend transarterial chemoembolization (TACE) as the treatment of choice in such cases, as this therapy can prolong survival. In such cases, international guidelines recommend transarterial chemoembolization (TACE) as the treatment of choice, as this therapy can prolong survival. TACE is a widely used interventional method in which a thin catheter is advanced to the liver artery supplying the tumor. Tiny beads loaded with a chemotherapeutic agent (doxorubicin) are then injected directly into the tumor nodules. The beads block the artery supplying the tumor, interrupting the blood supply to the tumor and causing it to die. In addition, the beads slowly release the chemotherapy drug doxorubicin into the tumor, which is intended to contribute to the complete death of the tumor cells. However, the studies also showed that complete death of the tumor node could only be achieved in approximately 25% of patients. The latest study results have revealed that one of the main causes of the incomplete response to TACE therapy is that cancer cells develop resistance to protect themselves against the chemotherapy drug doxorubicin. This resistance can be circumvented by inhibiting the enzyme ABCB1, allowing the chemotherapy drug to act on the tumor cells and kill them completely. The blood pressure medication nicardipine has a strong inhibitory effect on this enzyme. In this study, the investigators therefore want to investigate whether the response to TACE therapy can be improved by administering beads that release the active ingredient nicardipine in the tumor in addition to the chemotherapy drug doxorubicin, so that the tumor nodule cannot develop resistance and dies completely.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature,
* Age ≥18 years,
* Diagnosis of HCC by biopsy or by established imaging criteria using CT or MRI,
* At least one target lesion without prior treatment,
* Diameter of the target lesion ≥3 cm and ≤8 cm,
* Preserved liver function (no jaundice, no ascites, no overt hepatic encephalopathy).
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods for at least 3 months after the TACE treatment.

Exclusion Criteria:

* Any prior systemic therapy for advanced HCC,
* Diffuse tumor lesions, extrahepatic metastases, or vascular invasion,
* Hepatic encephalopathy,
* Uncontrolled ascites or pleural effusion,
* Jaundice,
* Severe hypotension or hemodynamic shock or need of vasoactive medications,
* Decompensated heart failure New York Heart Association (NYHA) class IV,
* eGFR < 15 mL/min/1.73 m2 per MDRD (Modification of Diet in Renal Disease) formula,
* Myocardial infarction within the last 6 months,
* Life expectancy <12 weeks,
* Contraindications to the class of drugs under study, e.g., known hypersensitivity or allergy to calcium antagonists,
* Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, etc. of the participant,
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within at least 3 months after the TACE treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
complete response rate (CRR) | 3 month
  of the target lesion at time point 3 months after TACE assessed by mRECIST (modified response evaluation criteria in solid tumors) in four-phase CT or contrast MRI according to standard liver imaging protocols
progression-free survival (PFS) | up to 12 month
  as defined as time to progression of any tumor treated as part of the trial or death of a patient.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 3 month
  Objective response (complete and partial) of the target lesion at time point 3 months assessed by mRECIST (modified response evaluation criteria in solid tumors).
Duration of response (DOR) | up to 12 month
Change in tumor markers | 3 and 6 month
Patient-reported outcomes | up to 1 year
  EuroQol 5-Dimension Questionnaire; 5-level version (EQ-5D-5L). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Overall survival | up to 12 month
Complete response of the target lesion | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Fahim Ebrahimi, PD Dr., Study Director — University Hospital, Basel, Switzerland
Locations (3):
- Switzerland (3):
  - University Hospital Basel, Basel
  - Hôpitaux Universitaires de Genève, Geneva
  - Kantonsspital St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: Undecided